CLINICAL TRIAL: NCT02047981
Title: Evaluating Impact of Azithromycin Mass Drug Administrations on All-cause Mortality and Antibiotic Resistance: Mortality Trial
Brief Title: Mortality Reduction After Oral Azithromycin: Mortality Study
Acronym: MORDORIMort
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Johns Hopkins University (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPP1032340-A
Record Dates: First submitted 2014-01-24; First posted 2014-01-29 (Estimated); Results first posted 2020-01-03 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Childhood Mortality
Keywords: Childhood mortality; Azithromycin; Mass treatment; Infection; Verbal Autopsy
MeSH Terms: conditions — Infections | interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Biannual mass oral azithromycin (Active Comparator): Comparison of childhood mortality in communities randomized to azithromycin versus communities randomized to placebo.
  Children aged 1 month to 60 months per community will be offered weight or height-based, directly observed, oral azithromycin suspension every 6 months for 2 years.
  In Niger during year 3, all communities will be offered azithroymcin.
  Interventions: Drug: Azithromycin
- Biannual mass oral placebo (Placebo Comparator): Comparison of childhood mortality in communities randomized to azithromycin versus communities randomized to placebo.
  Children aged 1 month to 60 months per community will be offered weight or height-based, directly observed, oral placebo every 6 months for 2 years
  In Niger during year 3, all communities will be offered azithroymcin.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Children aged 1 month to 60 months per community will be offered weight or height-based, directly observed, oral azithromycin suspension every 6 months for 2 years. In Niger during year 3, all communities will be offered azithroymcin.
  Other Names: Zithromax
  Arms: Biannual mass oral azithromycin
Drug: Placebo — Children aged 1 month to 60 months per community will be offered weight or height-based, directly observed, oral placebo every 6 months for 2 years. In Niger during year 3, all communities will be offered azithroymcin.
  Arms: Biannual mass oral placebo

SUMMARY:
Our long-term goal is to more precisely define the role of mass azithromycin treatments as an intervention for reducing childhood mortality. We propose a single multi-site (multi-country), cluster-randomized trial comparing communities randomized to oral azithromycin with those randomized to placebo. We hypothesize that mass azithromycin treatments will reduce childhood mortality.

DETAILED DESCRIPTION:
We will assess childhood mortality over three years, comparing communities where children aged 1-60 months receive biannual oral azithromycin ("Azithromycin" arm) for two years, to communities where the children receive biannual oral placebo ("Control" arm) for two years. During the third year at the Niger site only, everyone will receive azithromycin.

This is a cluster-randomized trial; at each site, communities within a contiguous area of 300,000 to 600,000 individuals will be randomized to azithromycin or placebo using simple random sampling.

Niger contingency study: In the event that mass distributions of oral azithromycin are proven to reduce mortality in 1-60 month-old children, then we will treat all communities in Niger with mass azithromycin distributions to test whether the intervention continues to reduce childhood mortality after the initial 2 years of mass treatments.

ELIGIBILITY:
Inclusion Criteria:

Communities

* The community location in target district.
* The community leader consents to participation in the trial
* The community's estimated population is between 200-2,000 people.
* The community is not in an urban area.

Individuals - All children aged 1-60 months (up to but not including the 5th birthday), as assessed via biannual census.

Exclusion Criteria:

Individuals

- Refusal of village chief (for village inclusion), or refusal of parent or guardian (for individual inclusion)

Ages: 1 Month to 60 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 190238 (Actual)
Dates: Start 2014-12; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom M Lietman, MD, Principal Investigator — University of California, San Francisco; Elodie J Lebas, RN, Study Director — University of California, San Francisco
Locations (6):
- United States (2):
  - UCSF Proctor Foundation, San Francisco, California
  - Johns Hopkins University, Baltimore, Maryland
- College of Medicine at the University of Malawi, Blantyre, Blantyre, Malawi
- The Carter Center, Niger, Niamey, Niger
- Kongwa Trachoma Project, Kongwa, Tanzania
- London School of Hygiene & Tropical Medicine, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hinterwirth A, Chen C, Yan D, Zhong L, Zhou Z, Liu Y, Keenan J, O'Brien KS, Lebas E, Porco TC, Lietman TM, Doan T. Co-selection of genetic antibiotic resistance in Streptococcus pneumoniae after repeated azithromycin mass drug administrations in Niger. Antimicrob Agents Chemother. 2025 Dec 23:e0156225. doi: 10.1128/aac.01562-25. Online ahead of print. PMID 41432154
- [Derived] Peterson B, Arzika AM, Amza A, Maliki R, Karamba AM, Moussa M, Kemago M, Liu Z, Houpt E, Liu J, Pholwat S, Doan T, Porco TC, Keenan JD, Lietman TM, O'Brien KS. Assessment of Spillover of Antimicrobial Resistance to Untreated Children 7-12 Years Old After Mass Drug Administration of Azithromycin for Child Survival in Niger: A Secondary Analysis of the MORDOR Cluster-Randomized Trial. Clin Infect Dis. 2024 Nov 22;79(5):1136-1143. doi: 10.1093/cid/ciae267. PMID 38739754
- [Derived] Arzika AM, Abdou A, Maliki R, Beido N, Kadri B, Harouna AN, Galo AN, Alio MK, Lebas E, Oldenburg CE, O'Brien KS, Chen C, Zhong L, Zhou Z, Yan D, Hinterwirth A, Keenan JD, Porco TC, Lietman TM, Doan T; MORDOR Study Group. Prolonged mass azithromycin distributions and macrolide resistance determinants among preschool children in Niger: A sub-study of a cluster-randomized trial (MORDOR). PLoS Med. 2024 May 6;21(5):e1004386. doi: 10.1371/journal.pmed.1004386. eCollection 2024 May. PMID 38709718
- [Derived] Chao DL, Arzika AM, Abdou A, Maliki R, Karamba A, Galo N, Beidi D, Harouna N, Abarchi M, Root E, Mishra A, Lebas E, Arnold BF, Oldenburg CE, Keenan JD, Lietman TM, O'Brien KS. Distance to Health Centers and Effectiveness of Azithromycin Mass Administration for Children in Niger: A Secondary Analysis of the MORDOR Cluster Randomized Trial. JAMA Netw Open. 2023 Dec 1;6(12):e2346840. doi: 10.1001/jamanetworkopen.2023.46840. PMID 38100110
- [Derived] Pickering H, Hart JD, Burr S, Stabler R, Maleta K, Kalua K, Bailey RL, Holland MJ. Impact of azithromycin mass drug administration on the antibiotic-resistant gut microbiome in children: a randomized, controlled trial. Gut Pathog. 2022 Jan 6;14(1):5. doi: 10.1186/s13099-021-00478-6. PMID 34991704
- [Derived] Arzika AM, Maliki R, Abdou A, Mankara AK, Harouna AN, Cook C, Hinterwirth A, Worden L, Zhong L, Chen C, Ruder K, Zhou Z, Lebas E, O'Brien KS, Oldenburg CE, Le V, Arnold BF, Porco TC, Keenan JD, Lietman TM, Doan T. Gut Resistome of Preschool Children After Prolonged Mass Azithromycin Distribution: A Cluster-randomized Trial. Clin Infect Dis. 2021 Oct 5;73(7):1292-1295. doi: 10.1093/cid/ciab485. PMID 34037753
- [Derived] Doan T, Worden L, Hinterwirth A, Arzika AM, Maliki R, Abdou A, Zhong L, Chen C, Cook C, Lebas E, O'Brien KS, Oldenburg CE, Chow ED, Porco TC, Lipsitch M, Keenan JD, Lietman TM. Macrolide and Nonmacrolide Resistance with Mass Azithromycin Distribution. N Engl J Med. 2020 Nov 12;383(20):1941-1950. doi: 10.1056/NEJMoa2002606. PMID 33176084
- [Derived] O'Brien KS, Arzika AM, Maliki R, Manzo F, Mamkara AK, Lebas E, Cook C, Bailey RL, West SK, Oldenburg CE, Porco TC, Arnold B, Keenan JD, Lietman TM; MORDOR Study Group. Biannual azithromycin distribution and child mortality among malnourished children: A subgroup analysis of the MORDOR cluster-randomized trial in Niger. PLoS Med. 2020 Sep 15;17(9):e1003285. doi: 10.1371/journal.pmed.1003285. eCollection 2020 Sep. PMID 32931496
- [Derived] Doan T, Hinterwirth A, Arzika AM, Worden L, Chen C, Zhong L, Oldenburg CE, Keenan JD, Lietman TM. Reduction of Coronavirus Burden With Mass Azithromycin Distribution. Clin Infect Dis. 2020 Nov 19;71(16):2282-2284. doi: 10.1093/cid/ciaa606. PMID 32426812
- [Derived] Keenan JD, Arzika AM, Maliki R, Elh Adamou S, Ibrahim F, Kiemago M, Galo NF, Lebas E, Cook C, Vanderschelden B, Bailey RL, West SK, Porco TC, Lietman TM; MORDOR-Niger Study Group. Cause-specific mortality of children younger than 5 years in communities receiving biannual mass azithromycin treatment in Niger: verbal autopsy results from a cluster-randomised controlled trial. Lancet Glob Health. 2020 Feb;8(2):e288-e295. doi: 10.1016/S2214-109X(19)30540-6. PMID 31981558
- [Derived] Bloch EM, Munoz B, Mrango Z, Weaver J, Mboera LEG, Lietman TM, Sullivan DJ Jr, West SK. The impact on malaria of biannual treatment with azithromycin in children age less than 5 years: a prospective study. Malar J. 2019 Aug 23;18(1):284. doi: 10.1186/s12936-019-2914-8. PMID 31443654
- [Derived] Doan T, Arzika AM, Hinterwirth A, Maliki R, Zhong L, Cummings S, Sarkar S, Chen C, Porco TC, Keenan JD, Lietman TM; MORDOR Study Group. Macrolide Resistance in MORDOR I - A Cluster-Randomized Trial in Niger. N Engl J Med. 2019 Jun 6;380(23):2271-2273. doi: 10.1056/NEJMc1901535. No abstract available. PMID 31167060
- [Derived] Keenan JD, Arzika AM, Maliki R, Boubacar N, Elh Adamou S, Moussa Ali M, Cook C, Lebas E, Lin Y, Ray KJ, O'Brien KS, Doan T, Oldenburg CE, Callahan EK, Emerson PM, Porco TC, Lietman TM. Longer-Term Assessment of Azithromycin for Reducing Childhood Mortality in Africa. N Engl J Med. 2019 Jun 6;380(23):2207-2214. doi: 10.1056/NEJMoa1817213. PMID 31167050
- [Derived] Porco TC, Hart J, Arzika AM, Weaver J, Kalua K, Mrango Z, Cotter SY, Stoller NE, O'Brien KS, Fry DM, Vanderschelden B, Oldenburg CE, West SK, Bailey RL, Keenan JD, Lietman TM; Macrolides Oraux pour Reduire les Deces avec un Oeil sur la Resistance (MORDOR) Study Group. Mass Oral Azithromycin for Childhood Mortality: Timing of Death After Distribution in the MORDOR Trial. Clin Infect Dis. 2019 May 30;68(12):2114-2116. doi: 10.1093/cid/ciy973. PMID 30561577
- [Derived] Keenan JD, Bailey RL, West SK, Arzika AM, Hart J, Weaver J, Kalua K, Mrango Z, Ray KJ, Cook C, Lebas E, O'Brien KS, Emerson PM, Porco TC, Lietman TM; MORDOR Study Group. Azithromycin to Reduce Childhood Mortality in Sub-Saharan Africa. N Engl J Med. 2018 Apr 26;378(17):1583-1592. doi: 10.1056/NEJMoa1715474. PMID 29694816
- [Derived] Porco TC, Stoller NE, Keenan JD, Bailey RL, Lietman TM. Public key cryptography for quality assurance in randomization for clinical trials. Contemp Clin Trials. 2015 May;42:167-8. doi: 10.1016/j.cct.2015.03.016. Epub 2015 Apr 7. No abstract available. PMID 25858004

RESULTS

PARTICIPANT FLOW:
Groups:
- Biannual Mass Oral Azithromycin: Comparison of childhood mortality in communities randomized to azithromycin versus communities randomized to placebo.
  Children aged 1 month to 60 months per community will be offered weight or height-based, directly observed, oral azithromycin suspension every 6 months for 2 years.
  In Niger during year 3, all communities will be offered azithroymcin.
  Azithromycin: Children aged 1 month to 60 months per community will be offered weight or height-based, directly observed, oral azithromycin suspension every 6 months for 2 years. In Niger during year 3, all communities will be offered azithroymcin.
- Biannual Mass Oral Placebo: Comparison of childhood mortality in communities randomized to azithromycin versus communities randomized to placebo.
  Children aged 1 month to 60 months per community will be offered weight or height-based, directly observed, oral placebo every 6 months for 2 years
  In Niger during year 3, all communities will be offered azithroymcin.
  Placebo: Children aged 1 month to 60 months per community will be offered weight or height-based, directly observed, oral placebo every 6 months for 2 years. In Niger during year 3, all communities will be offered azithroymcin.
Period: MORDOR Stage I Year 1-2
Arm/Group | Biannual Mass Oral Azithromycin | Biannual Mass Oral Placebo
Started | 97047 | 93191
Completed | 87650 | 84474
Not Completed | 9397 | 8717
Period: MORDOR Stage II Year 3
Arm/Group | Biannual Mass Oral Azithromycin | Biannual Mass Oral Placebo
Started | 37497 | 33294
Completed | 34611 | 30931
Not Completed | 2886 | 2363

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biannual Mass Oral Azithromycin | Biannual Mass Oral Placebo | Total
Number analyzed (Participants) | 97047 | 93191 | 190238
Age, Customized [Count of Participants; unit: Participants]
  Age group: 1-5 months | 7135 | 6870 | 14005
  Age group: 6-11 months | 12777 | 12318 | 25095
  Age group: 12-23 months | 18557 | 17886 | 36443
  Age group: 24-59 months | 58578 | 56117 | 114695
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47901 | 46019 | 93920
  Male | 49146 | 47172 | 96318
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 97047 | 93191 | 190238
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Niger | 40345 | 35747 | 76092
  Malawi | 39386 | 39534 | 78920
  Tanzania | 17316 | 17910 | 35226
Number of communities [Number; unit: communities] | 762 | 750 | 1512

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality Rate in Children Aged 1-60 Months
Description: This is a single multi-site trial, with each country as a secondary analysis. Also, an interim analysis of efficacy and futility will be conducted according to a pre-specified plan in the Statistical Analysis Plan.
Time Frame: 24 Months
Measure: Number; unit: deaths per 1000 person-years
Arm/Group | Biannual Mass Oral Azithromycin | Biannual Mass Oral Placebo
Number analyzed (Participants) | 97047 | 93191
deaths per 1000 person-years | 14.6 | 16.5

2. Primary Outcome: All-cause Mortality Rate in Children Aged 1-60 Months
Description: This was a pre-specified contingency study in Niger only in which all communities were treated with mass azithromycin during the third year of the study following the primary 24-month endpoint.
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: deaths per 1000 person-years
Arm/Group | Biannual Mass Oral Azithromycin | Biannual Mass Oral Placebo
Number analyzed (Participants) | 37497 | 33294
deaths per 1000 person-years | 23.3 [21.4 to 25.5] | 24.0 [22.1 to 26.3]

3. Secondary Outcome: Cause-specific Mortality Rate in Children Aged 1-60 Months, as Assessed From Verbal Autopsy (Niger Only)
Description: Deaths were assessed via biannual population census. A pre-specified outcome was cause of death, assessed by verbal autopsy.
Time Frame: 24 Months
Measure: Number (95% Confidence Interval); unit: Deaths per 1000 person years
Arm/Group | Biannual Mass Oral Azithromycin | Biannual Mass Oral Placebo
Number analyzed (Participants) | 40345 | 35747
Deaths per 1000 person years
  Injury | 0.22 [0.14 to 0.36] | 0.23 [0.14 to 0.38]
  Malnutrition | 0.39 [0.26 to 0.59] | 0.42 [0.28 to 0.63]
  AIDS | 0.12 [0.06 to 0.23] | 0.12 [0.06 to 0.24]
  Measles | 0.30 [0.19 to 0.46] | 0.28 [0.17 to 0.45]
  Meningitis | 0.82 [0.63 to 1.09] | 1.22 [0.96 to 1.57]
  Dysentery | 0.74 [0.55 to 0.98] | 1.14 [0.88 to 1.47]
  Diarrhea | 3.01 [2.59 to 3.49] | 3.60 [3.11 to 4.17]
  Pertussis | 0.04 [0.01 to 0.12] | 0.04 [0.01 to 0.14]
  Pneumonia | 3.27 [2.85 to 3.75] | 3.96 [3.46 to 4.53]
  Malaria | 5.60 [4.97 to 6.32] | 7.22 [6.43 to 8.11]
  Hemorrhagic fever | 0.08 [0.03 to 0.17] | 0.06 [0.02 to 0.16]
  Other infection | 4.24 [3.70 to 4.85] | 5.06 [4.44 to 5.78]
  Unspecified | 1.43 [1.17 to 1.75] | 1.81 [1.49 to 2.19]
  Total | 22.3 [20.9 to 23.9] | 27.3 [25.5 to 29.1]

4. Secondary Outcome: Cost-effectiveness of Mass Azithromycin Administration, Per Averted Childhood Death
Description: Cost-effectiveness of Mass Azithromycin Administration, Per Averted Childhood Death during the 24 month phase
Time Frame: 24 months
Population: all children 1-59 months treated
Measure: Mean (95% Confidence Interval); unit: usd per death averted
Arm/Group | Biannual Mass Oral Azithromycin | Biannual Mass Oral Placebo
Number analyzed (Participants) | 32369 | 32370
usd per death averted | 853 [581 to 1719] | 0 [0 to 0]

5. Secondary Outcome: All-cause and Cause-specific Health Clinic Visits in 1-60 Month-old Children
Description: We recorded clinic visits one year prior the study and during the first year of the study and collected outcomes of these visit.
Time Frame: 24 months
Population: Number of children visiting health centers
Measure: Number; unit: post-treatment clinical visits
Arm/Group | Biannual Mass Oral Azithromycin | Biannual Mass Oral Placebo
Number analyzed (Participants) | 12875 | 12809
post-treatment clinical visits | 5229 | 7647

6. Secondary Outcome: Cause-specific Mortality Rate in Children Aged 1-60 Months, as Assessed From Verbal Autopsy (Tanzania Only)
Description: At 6-monthly intervals a census of the communities was conducted, and for child deaths a verbal autopsy was performed to ascertain the cause using a standardized diagnostic classification. Mortality due to pneumonia or diarrhea by age group and arm are shown in the outcome measure data table below.
Time Frame: 24 Months
Measure: Number; unit: deaths per 100 person-years
Arm/Group | Biannual Mass Oral Azithromycin | Biannual Mass Oral Placebo
Number analyzed (Participants) | 17316 | 17910
deaths per 100 person-years
  Age group Mortality: 1- 5 months | 0.46 | 0.90
  Age group Mortality: 6- 11 months | 0.47 | 0.56
  Age group Mortality: 12 - 23 months | 0.29 | 0.29
  Age group Mortality: 24 - 59 months | 0.15 | 0.10

7. Secondary Outcome: Cause-specific Mortality Rate in Children Aged 1-60 Months, as Assessed From Verbal Autopsy (Malawi Only)
Description: Cause-specific mortality by intention-to-treat for the four main inferred causes of death in the study area.
Time Frame: 24 Months
Measure: Number (95% Confidence Interval); unit: deaths per 1000 person-years
Arm/Group | Biannual Mass Oral Azithromycin | Biannual Mass Oral Placebo
Number analyzed (Participants) | 39386 | 39534
deaths per 1000 person-years
  Pneumonia | 1.15 [0.92 to 1.44] | 1.40 [1.15 to 1.72]
  Malaria | 3.68 [3.25 to 4.17] | 3.84 [3.40 to 4.34]
  HIV/AIDS | 1.06 [0.84 to 1.34] | 1.54 [1.27 to 1.87]
  Diarrhoea | 0.67 [0.50 to 0.90] | 0.72 [0.54 to 0.95]

ADVERSE EVENTS:
Time Frame: 36 months.
Description: A SAE is any adverse event that:
  * Results in death
  * Is life-threatening (i.e., causes an immediate risk of death)
  * Requires inpatient hospitalization or prolongation of existing hospitalization
  * Results in persistent or significant disability or incapacity
  * Results in a congenital anomaly or birth defect
  Or that is considered to be:
  · An important medical event
  SAE reporting excludes mortality as measured for the primary outcome.
Arm/Group | Biannual Mass Oral Azithromycin | Biannual Mass Oral Placebo
All-Cause Mortality (participants affected / at risk) | 3262/97047 | 3392/93191
Serious Adverse Events (participants affected / at risk) | 3273/97047 | 3400/93191
Other Adverse Events (participants affected / at risk) | 0/97047 | 0/93191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biannual Mass Oral Azithromycin (N=97047) | Biannual Mass Oral Placebo (N=93191)
Suspected ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Suspected dehydration (General disorders) | 0 (0) | 2 (2)
Malaria (Infections and infestations) | 4 (4) | 3 (3)
Coma (General disorders) | 1 (1) | 0 (0)
ARI (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
(General disorders) | 4 (4) | 0 (0)
Death (General disorders) | 3262 (3262) | 3392 (3392)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/81/NCT02047981/Prot_001.pdf
  • Statistical Analysis Plan (2019-07-15): https://cdn.clinicaltrials.gov/large-docs/81/NCT02047981/SAP_000.pdf